CLINICAL TRIAL: NCT02358239
Title: Efficacy and Safety of Acupuncture for Dizziness and Vertigo in Emergency Department: a Clinical Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Po-Chi Hsu (Other)
Responsible Party: Sponsor-Investigator, Po-Chi Hsu, Ministry of Health and Welfare, Taiwan, Changhua Christian Hospital
Organization: Changhua Christian Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 120403
Record Dates: First submitted 2015-01-28; First posted 2015-02-06 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-02

CONDITIONS: Dizziness; Vertigo
Keywords: dizziness and vertigo; emergency department (ED); clinical trial; acupuncture
MeSH Terms: conditions — Dizziness; Vertigo; Emergencies | interventions — Acupuncture Therapy

ARMS (1):
- Efficacy and safety of acupuncture for dizziness and vertigo (Experimental): To evaluate the efficacy and safety of acupuncture in treating patients with dizziness and vertigo in ED.
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — Experiment group received acupuncture at Zusanli (ST36) and Neiguan (PC6) acupuncture points

SUMMARY:
Dizziness and vertigo account for roughly 4% of chief symptoms in the emergency department (ED). Pharmacological therapy is often solicited for these symptoms, such as vestibular suppressants, anti-emetics and benzodiazepines. However, every medication is accompanied with unavoidable side-effects. To the best of the investigators knowledge, no papers surveyed assess the feasibility of applying acupuncture as an emergent intervention means to the treatment of dizziness and vertigo. The investigators study targeted on filling in this gap by performing a clinical control trial to evaluate the efficacy and safety of traditional Chinese medicine - acupuncture - in treating patients with dizziness and vertigo in ED.

ELIGIBILITY:
Inclusion Criteria:

* Visit emergency department and stay in observation unit.
* Consult otolaryngologist and neurologist to rule in dizziness and giddiness, auditory vertigo, vertebrobasilar artery syndrome, and peripheral vestibular disorders - Ménière's disease, benign paroxymal peripheral vertigo, and vestibular neuritis.

Exclusion Criteria:

1. Serious comorbid conditions (for example, life-threatening condition or progressive central disorder).
2. Patients who cannot communicate reliably with the investigator or who are not likely to obey the instructions of the trial.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) of dizziness | after the first 30 minutes after acupuncture

REFERENCES:
- [Derived] Chiu CW, Lee TC, Hsu PC, Chen CY, Chang SC, Chiang JY, Lo LC. Efficacy and safety of acupuncture for dizziness and vertigo in emergency department: a pilot cohort study. BMC Complement Altern Med. 2015 Jun 9;15:173. doi: 10.1186/s12906-015-0704-6. PMID 26055400